CLINICAL TRIAL: NCT00430469
Title: Safety of a 0.5mg Dose of hLF1-11 Given for 10 Consecutive Days to Autologous Haematopoietic Stem Cell Transplant Recipients
Brief Title: Safety of hLF1-11 for the Treatment of Infectious Complications Among HSCT Recipients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Strategic company decision
Sponsor: AM-Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AMP 02-02; SC13; 2006-004012-52 (EudraCT Number)
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Fungal Infection; Bacterial Infection
Keywords: Lactoferrin; hLF; Neutropenia; Myeloablative; Treatment; Fungal; Bacterial; Infections; Bone marrow transplant
MeSH Terms: conditions — Mycoses; Bacterial Infections; Neutropenia; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: human lactoferrin (hLF1-11) — intravenous 0.5mg in NaCl-solution
  Other Names: hLF1-11

SUMMARY:
The safety and tolerability of hLF 1-11 given in multiple doses has to be established first in HSCT recipients who are at risk of developing, but have not yet developed, infectious complications due to invasive fungal or bacterial disease. These patients are different from healthy volunteers because they have received myeloablative treatment, which not only arrests haematopoiesis resulting in neutropenia but also induces mucosal barrier injury both of which predispose to infections, which typically occur during the week after transplant. It is therefore essential to know that hLF 1-11 is safe and well tolerated when given during neutropenia and mucosal barrier injury before infections ensue.

DETAILED DESCRIPTION:
Human lactoferrin (hLF) is a glycoprotein containing 692 amino acids and found in the saliva, milk, tears, and other body fluids. The peptide representing the first cationic domain, i.e. the peptide comprising the first eleven residues of hLF (further referred to as hLF1-11) was significantly more effective than the full length protein or the peptide representing the second cationic domain. As with other antimicrobial peptides, hLF1-11 shows poor antimicrobial activity under physiological conditions in vitro, but it is highly effective in vivo against infections due to a variety of microorganisms, including Gram negative and Gram positive bacteria and fungi. The objective is to develop hLF1-11 for the treatment of fungal and bacterial infections that develop during neutropenia that results from myeloablative therapy to prepare for a haematopoietic stem cell transplant(HSCT) formerly referred to as bone marrow transplant. Rates of infection and related morbidity are high in this population, making it an attractive target for testing clinically the proof-of-principle that hLF1-11 can provide effective treatment. Subsequently, hLF1-11 will be developed further as a systemic antifungal agent

ELIGIBILITY:
Inclusion Criteria:

Recipients will be eligible for inclusions if they satisfy the following conditions:

* Has been admitted for an autologous HSCT after myeloablative therapy with high-dose melphalan;
* Is being managed with a 3 or 4-lumen central venous catheter;
* Is at least 18 years old;
* Has a BMI <30 kg/M2;
* Has no medical reason for not participating
* Has adequate renal function (creatinine < 1.5 x ULN)
* Has adequate liver function (ASAT, ALAT < 2.5 x ULN, bilirubin < 1.5 x ULN);
* If a woman, is functionally post-menopausal
* Has not participated in a study of a new chemical molecular entity in the previous 3 months
* Is able and willing to participate;
* Has provided written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2009-03 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability as measured by adverse events, local tolerability, clinical chemistry, haematology, and vital signs | 28 Days

SECONDARY OUTCOMES:
Monitor for possible formation of hLF 1-11 specific antibodies. | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Donnelly, PhD, Principal Investigator — UMC St. Radboud Nijmegen
Locations (1):
- UMC St. Radboud, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Dijkshoorn L, Brouwer CP, Bogaards SJ, Nemec A, van den Broek PJ, Nibbering PH. The synthetic N-terminal peptide of human lactoferrin, hLF(1-11), is highly effective against experimental infection caused by multidrug-resistant Acinetobacter baumannii. Antimicrob Agents Chemother. 2004 Dec;48(12):4919-21. doi: 10.1128/AAC.48.12.4919-4921.2004. PMID 15561882
- [Background] Nibbering PH, Welling MM, Paulusma-Annema A, Brouwer CP, Lupetti A, Pauwels EK. 99mTc-Labeled UBI 29-41 peptide for monitoring the efficacy of antibacterial agents in mice infected with Staphylococcus aureus. J Nucl Med. 2004 Feb;45(2):321-6. PMID 14960656